CLINICAL TRIAL: NCT03073148
Title: Evaluation of Tangible Boost Replenishing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tangible Science (Industry)
Collaborators: University of Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 113133
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Contact Lens Solution
Keywords: Contact Lens Care Accessory

STUDY DESIGN:
Intervention Model Description: 2/3 of patients will be assigned to the Tangible Boost treatment arm of the study, and 1/3 of patients will be assigned to the placebo control arm.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tangible Boost (Experimental): Participants will treat their lenses with Tangible Boost after 30 days and again after 60 days.
  Interventions: Device: Tangible Boost
- Control (Placebo Comparator): Participants will treat their lenses with a placebo "Tangible Boost" kit containing saline after 30 days and again after 60 days.
  Interventions: Other: Placebo saline

INTERVENTIONS:
Device: Tangible Boost — Participants will treat their lenses with Tangible Boost, a kit designed to maintain the wettability of Hydra-PEG treated fluorosilicone acrylate lenses.
  Arms: Tangible Boost
Other: Placebo saline — Participants will treat their lenses with a placebo "Tangible Boost" kit, which contains saline in place of the Tangible Boost solution.
  Arms: Control

SUMMARY:
This study will evaluate Tangible Boost, a new contact lens care product which is designed to replenish the hydrogel layer on fluorosilicone acrylate lenses with Hydra-PEG. The Hydra-PEG coating is a poly(ethylene glycol)-based hydrogel that is covalently bound to the lens surface. This coating improves lens wettability, a common cause of patient discomfort. Tangible Boost is designed to maintain the wettability of Hydra-PEG lenses throughout the lens lifetime. Patients can use the Tangible Boost kit to reapply the Hydra-PEG coating each month at home.

ELIGIBILITY:
Inclusion Criteria:

* Habitual contact lens wear with a group 3 FDA approved rigid lens material, with 20-50% of subjects wearing corneal lenses
* Willing and able to sign the informed consent form
* 18 years or older

Exclusion Criteria:

* Eye injury or surgery within the 3 months immediately prior to enrollment for this trial
* Pre-existing ocular irritation that would preclude contact lens fitting
* Current enrollment in an ophthalmic clinical trial
* Evidence of systemic or ocular abnormality, infection, or disease which is likely to affect successful wear of contact lenses or use of the accessory solutions, as determined by the investigator
* Any use of medications for which contact lens wear could be contraindicated, as determined by the investigator
* Pregnant women and nursing mothers
* Visual acuity less than 20/20 when best corrected with contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria K Walker, OD MS, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

REFERENCES:
- See also: Tangible Science website — http://www.tangiblescience.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon enrollment in the study, patients received Hydra-PEG coated fluorosilicone acrylate RGP contact lenses. Assignment to the Tangible Boost or Control group occurred after 1 month of contact lens wear, on day 30. 4 participants that did not report back for visit 3 on day 30 were excluded from the study prior to assignment to a group.
Groups:
- Unassigned: Subjects that did not report back for visit 3 and were therefore not assigned to a treatment group.
Period: Overall Study
Arm/Group | Tangible Boost | Control | Unassigned
Started | 21 | 10 | 4
Completed | 21 | 10 | 0
Not Completed | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline measures are provided for all participants who were assigned to a study arm. Participants who dropped out of the study prior to assignment are not included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tangible Boost | Control | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (16) | 46 (16) | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 10 | 31
Corneal Staining [Median (Inter-Quartile Range); unit: units on a scale] — Corneal staining with lissamine green was used to identify damage to the corneal cells, which could have been caused by the contact lenses or treatments in the study. 5 regions in each eye were score on a scale of 0-4, resulting in a total possible range of 0-20. A higher score indicates more corneal damage. Left and right eye scores were averaged for each subject. Baseline data was collected after 1 month of lens wear in the study just prior to initial lens treatment with Tangible Boost or placebo control.
  units on a scale | 2.0 [0.25 to 3.75] | 2.0 [0 to 5.63] | 2.0 [0 to 4.5]
Visual Acuity (logMAR) [Median (Inter-Quartile Range); unit: units on a scale] — Visual acuity was calculated on a logMAR scale using high luminance, high contrast acuity charts. Baseline measurements were collected after 1 month of lens wear, prior to treatment with Tangible Boost or the placebo solution. A score of "0" indicates no vision loss, with higher scores indicating poorer vision.
  units on a scale | 0.11 [0.01 to 0.20] | 0.11 [-0.02 to 0.23] | 0.11 [0 to 0.20]
Non-invasive tear film break-up time [Mean (Standard Deviation); unit: seconds] — Tear break-up time was measured with the OCULUS Keratograph prior to lens treatment with Tangible Boost or the placebo, after 1 month of lens wear in the study.
  seconds | 17.40 (4.81) | 14.91 (6.48) | 16.59 (5.60)
Lens Fit [Count of Participants; unit: Participants] — Count of participants with acceptable lens fit (movement, centration, apical clearance, limbal clearance, and landing zone).
  Participants | 21 | 10 | 31
CLDEQ Score [Mean (Standard Deviation); unit: units on a scale] — The Contact Lens Dry Eye Questionnaire (CLDEQ) is used to evaluate the dry eye symptomology of contact lens wearers on a scale of 0-39. A lower score is indicative of greater comfort. Baseline measurements were collected prior to lens treatment after 1 month of lens wear.
  units on a scale | 16 (7) | 10 (8) | 14 (8)
Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The subjective comfort of lenses was evaluated on a scale of 1-100, with higher scores indicating better comfort.
  units on a scale | 64 (28) | 84 (22) | 73 (26)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Event Reports or Discontinuations
Description: A report of any adverse events or discontinuations that may have occurred. This measure includes adverse events unrelated to the treatment. See adverse events section for additional details.
Time Frame: Duration of study, 90 +/- 7 days after lens dispense visit.
Population: All subjects enrolled in the study were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Unassigned: Dropped out of study prior to assignment.
Arm/Group | Tangible Boost | Control | Unassigned
Number analyzed (Participants) | 21 | 10 | 4
Participants | 4 | 2 | 4

2. Primary Outcome: Corneal Staining
Description: Corneal staining with lissamine green was used to identify damage to the corneal cells, which may have been caused by the contact lenses or treatments in the study. 5 regions in each eye were scored on a scale of 0-4, resulting in a total possible range of 0-20. Left and right eye scores were averaged for each subject. A lower score indicates less corneal damage.
Time Frame: 1 day after treatment (day 31), final assessment (day 90)
Population: All participants that were assigned to a study arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 21 | 10
score on a scale
  1 day after treatment | 2.25 [.5 to 5.125] | 2.00 [.75 to 4.50]
  Final assessment | 1.5 [0 to 3.25] | 1.75 [0.75 to 4.375]
Statistical Analysis 1: Comparison: Tangible Boost; Test type: Equivalence — alpha = 0.05; p = 0.3577, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — alpha = 0.05; p = 0.9917, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment

3. Primary Outcome: Visual Acuity
Description: Visual acuity was calculated on a logMAR scale using high luminance, high contrast acuity charts. On the logMAR scale, a score of 0 indicates no vision loss, with higher scores indicating more vision loss.
Time Frame: 1 day after treatment (day 31), final assessment (day 90)
Population: All participants assigned to a study arm.
Measure: Median (Inter-Quartile Range); unit: logMAR visual acuity
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 21 | 10
logMAR visual acuity
  1 day after treatment | 0.12 [-.025 to 0.165] | 0.095 [-0.07 to 0.225]
  final assessment | 0.140 [0.020 to 0.225] | 0.060 [-0.0225 to 0.2725]
Statistical Analysis 1: Comparison: Tangible Boost; Test type: Equivalence — alpha = 0.05; p = 0.3239, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — alpha = 0.05; p = 0.8343, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment

4. Primary Outcome: Non-invasive Tear Film Break-up Time
Description: Tear break-up time was measured with the OCULUS Keratograph.
Time Frame: 1 day after treatment (day 31), final assessment (day 90)
Population: All participants that were assigned to a study arm. 1 participant was excluded due to malfunction of the keratograph during their visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 20 | 10
seconds
  1 day after treatment | 16.27 (4.32) | 19.84 (6.37)
  final assessment | 15.84 (4.64) | 18.30 (3.49)
Statistical Analysis 1: Comparison: Tangible Boost; Test type: Equivalence — alpha = 0.05; p = 0.4134, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — alpha = 0.05; p = 0.1192, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment

5. Primary Outcome: Number of Participants With Acceptable Lens Fit
Description: Count of participants with acceptable lens fit (movement, centration, apical clearance, limbal clearance, and landing zone).
Time Frame: final assessment (day 90)
Population: All participants that were assigned to a study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 21 | 10
Participants | 21 | 10

6. Secondary Outcome: CLDEQ Score
Description: The Contact Lens Dry Eye Questionnaire (CLDEQ) is used to evaluate the dry eye symptomology of contact lens wearers on a scale of 0-39. A lower score is indicative of greater comfort.
Time Frame: 1 day after treatment (day 31), final assessment (day 90)
Population: All participants that were assigned to a study group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 21 | 10
score on a scale
  1 day after treatment | 14.2 (8.9) | 7.9 (7.7)
  final assessment | 16.7 (8.0) | 11.4 (9.5)
Statistical Analysis 1: Comparison: Tangible Boost; Test type: Equivalence — alpha = 0.05; p = 0.1753, ANOVA — Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — alpha = 0.05; p = 0.1843, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment

7. Secondary Outcome: Visual Analog Scale (VAS)
Description: The subjective comfort of lenses was evaluated on a scale of 0-100, with higher scores indicating better comfort.
Time Frame: 1 day after treatment (day 31), final assessment (day 90)
Population: All participants that were assigned to a study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tangible Boost | Control
Number analyzed (Participants) | 21 | 10
score on a scale
  1 day after treatment | 78 (23) | 93 (9)
  final assessment | 75 (22) | 84 (20)
Statistical Analysis 1: Comparison: Tangible Boost; Test type: Equivalence — alpha = 0.05; p = 0.0765, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment
Statistical Analysis 2: Comparison: Control; Test type: Equivalence — alpha = 0.05; p = 0.1520, ANOVA; Repeated measures ANOVA comparing baseline, 1 day after treatment, and final assessment

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Tangible Boost | Control | Unassigned
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 4/21 | 2/10 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tangible Boost (N=21) | Control (N=10) | Unassigned (N=4)
Corneal Hydrops (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Mild, allergic-type reaction (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Acute inflammatory conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Mild conjunctival inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Preservative toxicity-type corneal sensitivity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Occurs in scleral lens wearers when preservatives remain in the lens bowl.
Contact lens associated red eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Decline in performance of the Hydra-PEG lenses was not observed in the control group; therefore, there was little opportunity to see improvements in outcome measures in the treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT03073148/Prot_SAP_ICF_000.pdf